CLINICAL TRIAL: NCT07148232
Title: Extended Intervention for Tobacco Use (EXIT) for People Experiencing Homelessness
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25632; NCI-2025-08620 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Cessation; Tobacco Abstinence; Tobacco Use; Tobacco Use Cessation; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use; Tobacco Use Disorder | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (extended intervention for tobacco use) (Experimental): Participants receive pharmacist provided one-time tobacco treatment using the five As: Ask, Advise, Assess, Assist and Arrange (5As) model and receives an initial monthly delivery of nicotine replacement therapy (NRT) for 3 months. Participants then receive the extended intervention for tobacco use (EXIT) that consists of: 1) health coach-delivered, weekly-to-monthly wellness-focused telephone coaching for 6 months addressing tobacco use within the context of co-occurring psychiatric and substance-use comorbidities and other life stressors, and 2) an additional session of pharmacist-delivered 5As with monthly delivery of NRT for an additional 6 months. Participants will provide CO samples for biochemical verification of smoking abstinence and complete questionnaires throughout the study.
  Interventions: Drug: Nicotine Replacement Therapy (NRT); Behavioral: Wellness Coaching
- Pharm-only (Other): Participants receive pharmacist provided one-time tobacco treatment using the 5As and receive monthly delivery of NRT for 3 months. Participants will provide CO samples for biochemical verification of smoking abstinence and complete questionnaires throughout the study.
  Interventions: Drug: Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Drug: Nicotine Replacement Therapy (NRT) — NRT will be administered as patch (transdermal), gum, or lozenge
  Other Names: NRT
Behavioral: Wellness Coaching — Delivered via phone call
  Arms: Treatment (extended intervention for tobacco use)

SUMMARY:
This study is investigating tobacco use and providing tobacco treatment among people experiencing homelessness in California, in San Francisco and Los Angeles.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Biochemically verified 7-day point prevalence tobacco abstinence at 6-months follow-up.

II. Use expired carbon monoxide (CO) to confirm self-reports of abstinence using a cut-off of CO ≤5 parts per million (ppm).

SECONDARY OBJECTIVES:

I. Biochemically-verified 7-day point prevalence tobacco abstinence at 3-months follow-up.

II. Measured at 6-months follow-up, a total number of expired carbon monoxide (CO-negative samples).

III. Measured at 6-months follow-up, longest duration of abstinence (i.e., total number of uninterrupted days abstinent), proportion with 50% reduction in expired CO for those who do not quit smoking.

IV. Use expired CO to confirm self-reports of abstinence using a cut-off of CO ≤5 ppm.

OUTLINE:

Participants will be randomized to one of two groups:

* Intervention group receives 6 months of pharmacist consultation, monthly delivery of nicotine replacement therapy, and telephone wellness coaching.
* Control group receives pharmacist consultation and monthly delivery of nicotine replacement therapy for 3 months.

Participants will be followed up at 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Ability of individual to understand a written informed consent document, and the willingness to sign it.
4. Staying at the recruitment site and meeting criteria for homelessness as defined by the Homeless Emergency and Rapid Transition to Housing Act.
5. Current smoking (smoking at least 5 cigarettes per day (cpd), verified via expired carbon monoxide (CO) >= 8 ppm using Micro+pro Smokerlyzer).
6. Having an intention to quit smoking within the next six months.
7. English speaking.

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.
2. Reasons that preclude the use of nicotine replacement therapy (NRT) (e.g., pregnancy or myocardial infarction in the past two weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who attended coaching sessions | up to 6 months
  The percentage of participants who attended at least 75% or 7 of the 14 coaching sessions will be reported.
Percentage of participants who used nicotine replacement therapy (NRT) | up to 6 months
  The percentage of participants who used at least 75% will adhere to using NRT for at least half of the treatment duration will be reported.
7-day point prevalence tobacco abstinence at month 6 | 6 months
  Biochemically verified 7-day point prevalence tobacco abstinence at 6-months follow-up will be reported.

SECONDARY OUTCOMES:
7-day point prevalence tobacco abstinence at month 3 | 3 months
  Biochemically verified 7-day point prevalence tobacco abstinence at 3-months follow-up will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Vijayaraghavan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No